CLINICAL TRIAL: NCT05122923
Title: Implementation of the S'TIM Serious-Game for Rehabilitation of Dysexecutive Disorders
Brief Title: Implementation of the S'TIM Serious-Game for Rehabilitation of Dysexecutive Disorders (S'TIM)
Acronym: S'TIM 1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-A00244-53
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Dysexecutive Syndrome; Serious Game

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Serious Game (Experimental)
  Interventions: Device: Serious Game S'TIM
- Patients without Serious Game (No Intervention)

INTERVENTIONS:
Device: Serious Game S'TIM — Video Game S'tim : the patient is inside a bedroom and he has to find a friend outside. this game will study the orientation, the memory of the patient
  Arms: Patients with Serious Game

SUMMARY:
This study proposes to improve the management of dysexecutive syndrome by a serious game (SG) in addition to the usual management including work in occupational therapy and neuropsychology.

ELIGIBILITY:
Inclusion Criteria:

* French-speaking male or female patient at least 18 years old
* Patient suffering from recent disorders (less than 6 months) of executive functions
* Patient with sufficient mobility of the upper limb (mobility of the dominant upper limb greater than 70 °) to interact with the device.
* Patient affiliated or beneficiary of a social security scheme
* Patient having signed the free and informed consent.

Exclusion Criteria:

* Patient participating in another clinical study
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision,
* Pregnant or breastfeeding woman,
* Patient hospitalized without consent.
* Patient with unstable psychiatric disorders
* Patient with comprehension disorders (alexia, visual agnosia, illiteracy, not understanding the language, etc.)
* Patient with executive function disorders greater than 6 months
* Negligent hemi patient
* Patient not familiar with the French language
* Patient with major neuro-visual disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-12-03 (Estimated); Study Completion 2022-06-03 (Estimated)

PRIMARY OUTCOMES:
The effect of using the serious-game S'TIM in terms of cognition | 6 weeks
  TAP sub-test ERFC : overall cognitive functions BREF : presence or absence of a cognitive and / or behavioral dysexecutive syndrome
The effect of using the serious-game S'TIM at 6 weeks in terms of metacognition with the BRIEF-A | 6 weeks
  Behaviour Rating Inventory of Executive Function, Adult
The effect of using the serious-game S'TIM at 6 weeks in terms of behavior with BRIEF-A | 6 weeks
  Behaviour Rating Inventory of Executive Function, Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de Provence Bourbonne, Aubagne, France